CLINICAL TRIAL: NCT00005973
Title: Phase I Study of Farnesyl Transferase Inhibitor BMS-214662 (NSC 710086D) in Solid Tumors
Brief Title: BMS-214662 in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02343; ID99-304; U01CA062461 (NIH); CDR0000067960 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — 7-cyano-2,3,4,5-tetrahydro-1-(1H-imidazol-4-ylmethyl)-3-(phenylmethyl)-4-(2-thienylsulfonyl)-1H-1,4-benzodiazepine

ARMS (1):
- Treatment (Experimental): Patients receive BMS-214662 IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BMS-214662; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: BMS-214662 — Given IV
  Other Names: farnesyltransferase inhibitor BMS-214662; FTI BMS 214662
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of BMS-214662 in treating patients who have solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of BMS-214662 in patients with solid tumors.

II. Evaluate intermediate biological endpoints as surrogates for the effectiveness of this drug in these patients.

III. Determine the nature of dose limiting toxicity of this drug in this patient population.

IV. Determine the recommended phase II regimen of this drug in these patients. V. Establish a pharmacologic and pharmacokinetic profile of this drug in these patients.

OUTLINE: This is a dose escalation study.

Patients receive BMS-214662 IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-214662 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicities.

Patients are followed every 3 months for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant solid tumor for which a standard curative therapy does not exist
* Performance status - Karnofsky 70-100%
* At least 6 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 2 times upper limit of normal
* Albumin at least 3.0 g/dL
* Creatinine no greater than 1.5 mg/dL
* No uncontrolled heart disease
* No history of clinically significant cardiac arrhythmia that could be exacerbated by QT interval prolongation
* Corrected QT interval no greater than 450 milliseconds
* Must not require total parenteral nutrition
* No manifestations of malabsorption syndrome due to prior surgery, gastrointestinal disease, or unknown reasons
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No signs or symptoms of acute infection requiring systemic therapy
* No grade 3 or 4 neurotoxicity from prior anticancer treatment or neuropathy from any cause
* No confusion, disorientation, or psychiatric illness that may preclude study
* No more than 3 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas or mitomycin) and recovered
* No other concurrent antineoplastic agents
* No concurrent hormonal anticancer therapy
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* Prior drugs known to prolong the QT interval allowed if they can be safely discontinued for a time period equal to 4 elimination half-lives prior to administering study drug
* No drugs known to prolong the QT interval during and for 24 hours after study drug
* No concurrent therapy with known CYP3A4 substrates
* No other concurrent investigational agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-04; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the dose level among the 9 levels studied having toxicity rate closest to a target of 33%, graded according to CTC version 2.0 | Up to 6 weeks
  Toxicity is defined as grade 3, 4 non-hematologic and grade 4 hematologic (neutropenia and thrombocytopenia) toxicity. The continual reassessment method (CRM) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States